CLINICAL TRIAL: NCT05307692
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind Study to Investigate the Safety, Tolerability, and Clinical Efficacy of Seltorexant (JNJ-42847922) on Behavioral and Psychological Symptoms of Dementia in Patients With Probable Alzheimer's Disease
Brief Title: A Study of Seltorexant in Participants With Probable Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109177; 42847922ALZ2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-03-25; First posted 2022-04-01 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — seltorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Seltorexant (Experimental): Participants will receive single oral dose of seltorexant 20 milligrams (mg) tablet once daily from Day 1 to Day 42.
  Interventions: Drug: Seltorexant
- Placebo (Placebo Comparator): Participants will receive single oral dose of matching placebo tablet once daily from Day 1 to Day 42.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Seltorexant — Seltorexant 20 mg will be administered orally as a tablet.
  Other Names: JNJ-42847922
  Arms: Seltorexant
Drug: Placebo — Matching placebo will be administered orally as a tablet.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of seltorexant versus placebo on the sum of Agitation and Aggression domain scores (A plus A) of the Neuropsychiatric Inventory-Clinician rating (NPI-C) in participants with probable Alzheimer's Disease (AD) with clinically significant agitation/aggression.

ELIGIBILITY:
Inclusion Criteria:

* Participant has received a diagnosis of probable Alzheimer Disease (AD) (Diagnostic and Statistical Manual of Mental Disorders-5 [DSM-5]) with the following characteristics at screening: Clinical Dementia Rating (CDR) global score greater than or equal to (>=) 1; Mini-Mental State Examination (MMSE) total score of 10 to 24 (inclusive)
* Participant meets the criteria of a syndrome diagnosis of agitation based on International Psychogeriatric Association (IPA) consensus clinical and research definition of agitation in cognitive disorders for at least 2 weeks before screening
* Participant meets the criteria of Neuropsychiatric Inventory (NPI-12) Agitation/Aggression (A/A) domain score >= 4 with frequency score >= 2 at screening and baseline with no more than 35 percent (%) of improvement in NPI-12 A/A domain score from the screening to baseline assessments
* Female participants must be postmenopausal before study entry (amenorrhea for at least 12 months)
* Body Mass Index (BMI) within the range 18-40 kilograms per square meter (kg/m^2) (inclusive)

Exclusion Criteria:

* Participant fulfils diagnostic criteria for non-Alzheimer's Dementia: example, Frontotemporal Dementia (FTD), Diffuse Lewy Body Dementia (DLBD), and post-stroke dementia, based on clinical history. (Participants may be included with mixed AD/vascular dementia)
* Participant has a clinically significant acute illness within 7 days prior to study intervention administration
* Participants with a history of delirium within 30 days prior to or during screening
* Participant with a cause of agitation that is not secondary to dementia (such as pain) or significant history of aggression prior to dementia based on investigator judgment
* Participants who are not stable on concomitant medications or take prohibited medications

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research and Development, LLC Clinical Trial, Study Director — Janssen Research and Development LLC
Locations (25):
- United States (25):
  - Medical Advancement Center of Arizona, Tempe, Arizona
  - Sunwise Clinical Research, Lafayette, California
  - Luminous Clinical Research, Homestead, Florida
  - Global Medical Institutes, Miami, Florida
  - Office of Emilio Mantero-Atienza, MD, Miami, Florida
  - Allied Biomedical Research Institute (ABRI), Inc, Miami, Florida
  - Quantix Research, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Florida International Research Center (FIRC), Miami, Florida
  - P&S Research, LLC, Miami, Florida
  - IMIC Inc, Miami, Florida
  - Biovision Medical, Miami, Florida
  - South Florida Research Center Inc., Miami Springs, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Accel Clinical Research, Seminole, Florida
  - Sonar Clinical Research, Atlanta, Georgia
  - NeuroTrials Research Inc, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Ochsner Medical Center, New Orleans, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Richmond Behavioral Associates, Staten Island, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Gill Neuroscience, Cypress, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Memory Clinic Inc, Bennington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- DB: Placebo: Participants received placebo matching to seltorexant tablet orally once daily at bedtime from Day 1 to Day 42.
- DB: Seltorexant: Participants received seltorexant 20 milligrams (mg) orally once daily at bedtime from Day 1 to Day 42.
- Follow-up (FU): Placebo; FU: Seltorexant: After the completion of double-blind phase, participants entered the post-treatment follow up phase and were followed up until Day 57.
Period: Double-blind (DB) Phase (Day 1- Day 43):
Arm/Group | DB: Placebo | DB: Seltorexant | Follow-up (FU): Placebo | FU: Seltorexant
Started | 44 | 44 | 0 | 0
Treated | 42 | 43 | 0 | 0
Completed | 39 | 35 | 0 | 0
Not Completed | 5 | 9 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Protocol-specified withdrawal criterion met | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0
Not completed — Randomized but not treated | 2 | 1 | 0 | 0
Period: FU Phase (Day 43 to Day 57):
Arm/Group | DB: Placebo | DB: Seltorexant | Follow-up (FU): Placebo | FU: Seltorexant
Started | 0 | 0 | 39 | 38 (Three participants, who discontinued treatment during the DB phase (and so did not complete DB). They continued and entered the follow up phase.)
Completed | 0 | 0 | 39 | 34
Not Completed | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants who took at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | DB: Placebo | DB: Seltorexant | Total
Number analyzed (Participants) | 42 | 43 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (7.75) | 73.4 (6.18) | 73 (6.97)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 7 | 2 | 9
  From 65 to 84 years | 35 | 40 | 75
  85 years and over | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 54
  Male | 16 | 15 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 43 | 82
  Not Hispanic or Latino | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 37 | 41 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 42 | 43 | 85
Age Categorical [Count of Participants; unit: Participants]
  Adults (18-64 years) | 7 | 2 | 9
  From 65 to 84 years | 35 | 40 | 75
  85 years and over | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Neuropsychiatric Inventory Clinician Version (NPI-C) Sum of Agitation and Aggression Domain Scores (NPI-C A+A) at Day 43: Analyzed Under Estimand 1
Description: The NPI-12, measure of psychobehavioral disturbances assessed frequency and severity of disturbances in 12 domains, based on a caregiver interview. Frequency for each domain was rated on a 4-point scale (from 1=rarely to 4=very often) and severity on a 3-point scale (from 1=mild to 3=severe), with the score for each domain being product of frequency and severity scores, such that each domain was scored from 1 to 12. The NPI-12 total score was the sum of 12 domain scores, ranging from 0 (best) to 144 (worst), higher score represented greater frequency and worst severity of the symptoms. NPI-C was an instrument developed on basis of original NPI that gives a score based on product of frequency and severity ratings of 12 symptom domains that were summed to a total score. NPI-C domains: agitation and aggression NPI-C A+A were scored based on both caregiver and participant interviews and score ranged from 0 (does not occur) to 63 (severe). Higher scores indicated more severity.
Time Frame: Baseline (Day 1) and Day 43
Population: Full analysis set (FAS) included all randomized participants who took at least 1 dose of study intervention. 'N' (number of participants analyzed): participants evaluable for this outcome measure. Estimand 1 used to analyze benefit from seltorexant 20 mg versus placebo in adults and elderly participants with probable Alzheimer's disease (AD) with clinically significant agitation/aggression who took study intervention as directed and regardless treatment discontinuation without treatment switch.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | DB: Placebo | DB: Seltorexant
Number analyzed (Participants) | 37 | 36
Score on a scale | -9.6 (8.35) | -13.4 (9.31)
Statistical Analysis 1: Comparison: DB: Placebo vs DB: Seltorexant; Test type: Superiority; p = 0.308, Mixed model repeated measures; Difference of Least Square (LS) Means = -1.5, 80% CI 2-sided [-3.41 to 0.39], Standard Error of Mean 1.47

2. Primary Outcome: Change From Baseline in NPI-C A+A at Day 43: Analyzed Under Estimand 2
Description: The NPI-12, measure of psychobehavioral disturbances assessed frequency and severity of disturbances in 12 domains, based on a caregiver interview. Frequency for each domain was rated on a 4-point scale (from 1=rarely to 4=very often) and severity on a 3-point scale (from 1=mild to 3=severe), with the score for each domain being product of frequency and severity scores, such that each domain was scored from 1 to 12. The NPI-12 total score was the sum of 12 domain scores, ranging from 0 (best) to 144 (worst), higher score represented greater frequency and worst severity of the symptoms. NPI-C was an instrument developed on the basis of original NPI that gives a score based on product of frequency and severity ratings of 12 symptom domains that were summed to a total score. NPI-C domains: agitation and aggression NPI-C A+A were scored based on both caregiver and participant interviews and score ranged from 0 (does not occur) to 63 (severe). Higher scores indicated more severity.
Time Frame: Baseline (Day 1) and Day 43
Population: Full analysis set (FAS) included all randomized participants who took at least 1 dose of study intervention. 'N' (number of participants analyzed): participants evaluable for this outcome measure. Estimand 2 was used to analyze benefit from seltorexant 20 mg versus placebo in adults and elderly participants with probable AD with clinically significant agitation/aggression who took study intervention as directed and regardless of treatment discontinuation without treatment switch.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | DB: Placebo | DB: Seltorexant
Number analyzed (Participants) | 38 | 36
Score on a scale | -9.6 (8.25) | -13.4 (9.31)
Statistical Analysis 1: Comparison: DB: Placebo vs DB: Seltorexant; Test type: Superiority; p = 0.282, Mixed model repeated measures; Difference of Least Square (LS) Means = -1.5, 80% CI 2-sided [-3.33 to 0.29], Standard Error of Mean 1.42

3. Secondary Outcome: Change From Baseline in Cohen-Mansfield Agitation Inventory- Community Version (CMAI-C) Total Score at Day 43
Description: The CMAI-C, 37-item scale, measured the ability of a drug to reduce overall frequency of agitation symptoms, including aggressive behaviors. Individual items were rated by the clinician on a scale of 1 (never) to 7 (several times per hour) in which higher score represented the most frequent for each item assessed. CMAI-C total score was a sum of all categories that ranged from 37 (never) to 259 (several times), where higher score indicated greater severity.
Time Frame: Baseline (Day 1) and Day 43
Population: FAS included all randomized participants who took at least 1 dose of study intervention. Here, 'N' (overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | DB: Placebo | DB: Seltorexant
Number analyzed (Participants) | 38 | 36
Score on a scale | -17.5 (18.67) | -20.3 (21.69)

4. Secondary Outcome: Change From Baseline in Sleep Disorder Inventory (SDI) Average Total Score at Day 43
Description: SDI: based on caregiver (CG) interview and expanded version of item 11 (night-time behavioral disturbances) of NPI-12. It described frequency, severity and CG burden of sleep-disturbed behaviors for period prior to its administration. It consisted of 7 sub-questions from NPI-12 sleep disturbance item. Each sub-question was made into separate questions with frequency, severity, and CG distress rated with respect to participant. SDI score derived after CG rated frequency, severity of each of 7 separate sleep disturbance symptoms. CG distress ratings were not part of SDI total score, but distress was measured. Frequency scored on scale of 0 (not present) to 4 (once or more per day), severity scored on scale of 0 (not present) to 3 (occurrence of nighttime behaviors) and CG distress rated on scale of 0 (not at all) to 5 (extremely). SDI average total score=average frequency of item 1 to 7 multiplied with average severity of items 1 to 7; ranged from 0 to 12; higher score=greater severity.
Time Frame: Baseline and Day 43
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | DB: Placebo | DB: Seltorexant
Number analyzed (Participants) | 36 | 36
Score on a scale | -0.8 (1.02) | -0.5 (0.90)

5. Secondary Outcome: Observed Plasma Concentrations of Seltorexant and Its Metabolite (M12)
Description: The pharmacokinetic (PK) sample collection was done based on the availability of the participants either on Day 15 or 43 and thus collected data were analyzed and summary data were reported in this outcome measure. Plasma samples were analyzed using liquid chromatography/mass spectrometry/mass spectrometry (LC-MS/MS) method.
Time Frame: Either Day 15 (8 and 14 hours post dose on night of Day 14) or Day 43 (8 and 14 hours post dose on night of Day 42)
Population: The PK analysis set included all randomized participants to the seltorexant treatment group and with at least one PK sample taken. Here, 'N' (overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | DB: Seltorexant
Number analyzed (Participants) | 22
nanograms per milliliter (ng/mL)
  Total Seltorexant | 121 (156)
  Total M12 | 141 (164)

ADVERSE EVENTS:
Time Frame: Double-blind (DB) Phase: From Day 1 up to Day 43; Follow up Phase: From Day 44 to Day 57
Description: All-cause mortality was anlyzed on all randomized participants. Serious adverse events and other adverse events were analyzed on safety analysis set which included all randomized participants who took at least 1 dose of study intervention.
Arm/Group | DB: Placebo | DB: Seltorexant | Follow-up (FU): Placebo | FU: Seltorexant
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44 | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/42 | 1/43 | 0/39 | 1/38
Other Adverse Events (participants affected / at risk) | 4/42 | 6/43 | 0/39 | 2/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Placebo (N=42) | DB: Seltorexant (N=43) | Follow-up (FU): Placebo (N=39) | FU: Seltorexant (N=38)
Pancreatic Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Placebo (N=42) | DB: Seltorexant (N=43) | Follow-up (FU): Placebo (N=39) | FU: Seltorexant (N=38)
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0
Supraventricular Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Malignant Biliary Obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Tension Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Abnormal Dreams (Psychiatric disorders) | 0 | 1 | 0 | 0
Confusional Arousal (Psychiatric disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-04-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT05307692/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT05307692/SAP_001.pdf